CLINICAL TRIAL: NCT07379463
Title: Amino Acid Transporter System PET/CT Imaging in AATS-Related Diseases
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Shaobo Yao, PhD, Prof., Tianjin Medical University
Other Study IDs: TJMUGH-14
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Amino-Acid Transport Disorder; Primary Hyperparathyroidism; Glioma
Keywords: PET/CT; Amino acid transporter; MET; FET
MeSH Terms: conditions — Hyperparathyroidism, Primary; Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment: Each subject receive a single intravenous injection of 11C/18F-MET/FET, and undergo PET/CT imaging within the specificed time.
  Interventions: Diagnostic Test: 11C/18F-MET/FET

INTERVENTIONS:
Diagnostic Test: 11C/18F-MET/FET — Each subject receive a single intravenous injection of 11C/18F-MET/FET, and undergo PET/CT imaging within the specificed time

SUMMARY:
To evaluate the potential usefulness of 11C/18F-MET/FET positron emission tomography/ computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various amino acid transporter system (AATS)-related disease patients.

DETAILED DESCRIPTION:
Subjects with various AATS-related disease (Primary Hyperparathyroidism, Glioma, et al) patients underwent 11C/18F-MET/FET PET/CT either for an initial assessment or for recurrence detection. Lesions uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 11C/18F-MET/FET were calculated.

ELIGIBILITY:
Inclusion Criteria:

1. adult patients (aged 18 years or order);
2. patients with suspected or newly diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report);
3. patients who had scheduled AATS PET/CT scan;
4. patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

1. patients with non-malignant lesions;
2. patients with pregnancy;
3. the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. adult patients (aged 18 years or order);
  2. patients with suspected or newly diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report);
  3. patients who had scheduled AATS PET/CT scan;
  4. patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-08-29 (Actual); Primary Completion 2033-08-29 (Estimated); Study Completion 2033-08-29 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of AATS for each target lesion of subject or suspected primary tumor or/and metastasis.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity and accuracy of AATS PET/CT were calculated.

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No